CLINICAL TRIAL: NCT00590759
Title: A Clinical Evaluation of the GORE TAG Thoracic Endoprosthesis in the Primary Treatment of Descending Thoracic Aortic Aneurysms
Brief Title: Evaluation of the GORE TAG Thoracic Endoprosthesis in the Treatment of Aneurysms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAG 05-02
Record Dates: First submitted 2007-12-20; First posted 2008-01-11 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GORE TAG® Thoracic Endoprosthesis (Other)
  Interventions: Device: GORE TAG® Thoracic Endoprosthesis

INTERVENTIONS:
Device: GORE TAG® Thoracic Endoprosthesis — implant

SUMMARY:
The purpose of this post-approval study is to evaluate the long-term performance of the GORE TAG® Thoracic Endoprosthesis (TAG device) in the primary treatment of descending thoracic aortic (DTA) aneurysms

ELIGIBILITY:
Inclusion Criteria:

1. Descending thoracic aortic aneurysm deemed to warrant surgical repair:

   1. Fusiform aneurysm greater than or equal to 2 times diameter of normal adjacent aorta
   2. Saccular aneurysm
2. Anatomy meets GORE TAG Thoracic Endoprosthesis specification criteria as indicated in the Instructions for Use (Appendix A)
3. Minimum 2 cm non-aneurysmal segment proximal and distal to the aneurysm

   • <60 degree angle in the aortic arch may require additional length of non-aneurysmal segment if the arch is included in the treatment segment
4. Life expectancy > 2 years
5. Surgical Candidate

   * ASA Class I, II, III, or IV
   * NYHA Class I, II, III or no heart disease
6. Male or infertile female
7. Minimum 21 years of age
8. Able to comply with protocol requirements
9. Signed Informed Consent Form

Exclusion Criteria:

1. 4 mm aortic taper and inability to use devices of different diameters, to compensate for the taper, in the treatment area of the aorta
2. Significant thrombus at the proximal or distal implantation zones
3. Mycotic aneurysm
4. Hemodynamically unstable aneurysm rupture (non-contained aneurysm rupture)
5. Acute or chronic aortic dissection
6. Planned occlusion of the left carotid or celiac arteries
7. "Planned" concomitant surgical procedure (other than left subclavian transposition) or previous major surgery within 30 days
8. Myocardial infarction or cerebral vascular accident within 6 weeks
9. Severe respiratory insufficiency sufficient that precludes open thoracotomy
10. Renal insufficiency (Creatinine > 2.0 mg/dL) with or without dialysis
11. Degenerative connective tissue disease, e.g., Marfan or Ehler-Danlos Syndrome
12. Participation in another investigational device or drug study within 1 year
13. Documented history of drug abuse within 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Morasch, M.D., Principal Investigator — St. Vincent's Healthcare, Billings MT
Locations (25):
- United States (25):
  - Phoenix, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Greeley, Colorado
  - Gainesville, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Peoria, Illinois
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - St Louis, Missouri
  - Albany, New York
  - New York, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Seattle, Washington
  - Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Thoracic Endograft: GORE TAG® Thoracic Endoprosthesis: implant
Period: Overall Study
Arm/Group | Thoracic Endograft
Started | 150
Completed | 70
Not Completed | 80
Not completed — Death | 52
Not completed — Lost to Follow-up | 28

BASELINE CHARACTERISTICS:
Arm/Group | Thoracic Endograft
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 102
Region of Enrollment [Number; unit: participants]
  United States | 150

OUTCOME MEASURES:

1. Primary Outcome: Aneurysm Related Death
Description: Freedom from aneurysm related mortality for TAG 05-02 subjects
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Thoracic Endograft
Number analyzed (Participants) | 150
participants | 4

2. Secondary Outcome: A Subset of Major Adverse Events Will be Evaluated in Subjects Treated With the TAG Device and Subjects Treated With Open Surgical Repair.
Description: Proportion of subjects in TAG 05-02 with MAEs
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Thoracic Endograft
Number analyzed (Participants) | 150
participants | 22

ADVERSE EVENTS:
Time Frame: Total Study Follow-up.
Description: Note - the severity of adverse events (serious vs non-serious) was not collected, so all events, regardless of whether they would be classified as serious or not, are reported under "Other adverse events"
Arm/Group | 0502 TAG Device Subjects
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 147/150
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0502 TAG Device Subjects (N=150)
Bleeding Complication (Blood and lymphatic system disorders) | 52
Cardiac Complication (Cardiac disorders) | 64
Bowel Complication (Gastrointestinal disorders) | 54
Additional Implantation (General disorders) | 16
Other Complication (General disorders) | 102
Endoleak (Injury, poisoning and procedural complications) | 58
Wound Complication (Injury, poisoning and procedural complications) | 43
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15
Neurologic Complication (Nervous system disorders) | 62
Genitourinary (Renal and urinary disorders) | 40
Renal Function Complication (Renal and urinary disorders) | 26
Pulmonary Complication (Respiratory, thoracic and mediastinal disorders) | 67
Vascular Complication (Vascular disorders) | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Gore has the right to review disclosures, requesting a delay of less than 90 days. Each investigator will postpone single center publications until after disclosure of multi-center data, less than 12 months from study completion/termination at all participating sites